CLINICAL TRIAL: NCT07211581
Title: Predicting Factors of Post-Total Thyroidectomy Hypocaӏcemia
Status: Completed | Type: Observational
Sponsor: Al Safwa University College (Other)
Responsible Party: Principal Investigator, Mohammed AbdulZahra Sasaa, Predicting Factors of Post-Total Thyroidectomy Hypocaӏcemia, Al Safwa University College
Other Study IDs: AlSafwaUC
Record Dates: First submitted 2025-09-17; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Hypocalcemia After Total Thyroidectomy
Keywords: Predicting Factors.; Total Thyroidectomy.; Hypocalcemia
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: total thyroidectomy — both lobes removed and observe the calcemic level

SUMMARY:
Predicting post-total thyroidectomy hypocalcemia involves a combination of patient-specific, disease-related, and surgical factors. Key predictive factors include the intrinsic characteristics of the thyroid disease, pre-operative levels of calcium and vitamin D, the degree of parathyroid gland manipulation or injury, advanced age, and pre-existing hyperthyroidism. While no single factor is definitive, a low post-operative parathyroid hormone (iPTH) level is a strong indicator of developing hypocalcemia

ELIGIBILITY:
Inclusion Criteria:

1. patients requiring total thyroidectomy.
2. age between 18-75 years old
3. both gender
4. no co-existing disease.

Exclusion Criteria:

1. previous hemithyroidectomy, lobectomy, resection of the parathyroid gland. 2. 2. patients with missing laboratory data, previous subtotal thyroidectomy.

3. diagnosed pathology of the parathyroid gland

Ages: 21 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 123 patients who underwent total thyroidectomy for various thyroid diseases were included in the study, performed by a group of surgeons.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
hypocalcemia incidence | 1 day and 2 weeks after surgery
hypocalcemia other factors related to clinical status. | 1 day and 2 weeks after surgery
  Comparison of Serum Calcium levels of the studied group reported Comparison of PTH levels between hypocaӏcemia and Eucalcemic

CONTACTS AND LOCATIONS:
Overall Officials: 1. Ali Fadhil Zaidan, PhD, Study Chair — mustaqbal university
Locations (1):
- Mustaqbal University, Sfax, Safx, Tunisia

IPD SHARING:
Plan to Share IPD: No